CLINICAL TRIAL: NCT01206205
Title: IFM2008: Frontline Therapy in de Novo Multiple Myeloma Patients Under 65, (a Phase 2 Multicenter Trial)
Brief Title: Frontline Therapy in de Novo Multiple Myeloma Patients Under 65
Acronym: IFM2008
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Celgene Corporation (Industry); Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0805603
Record Dates: First submitted 2010-09-17; First posted 2010-09-21 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma
Keywords: De novo Multiple Myeloma; Bortezomib; Lenalidomide; induction therapy; consolidation therapy; maintenance therapy; High dose therapy; frontline therapy including new drugs and high dose therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide, Bortezomib (Experimental): 3 induction cycles of bortezomib, lenalidomide and dexamethasone (VRD) followed by high dose melphalan and autologous stem cell transplantation.
  Two months after haematological recovery, patients will receive 2 consolidation cycles of VRD and maintenance therapy for 1 year with lenalidomide.
  Interventions: Drug: Lenalidomide, Bortezomib

INTERVENTIONS:
Drug: Lenalidomide, Bortezomib — Induction:
  3 cycles of 21 days of Dexamethasone : 40 mg/j, days 1, 8 et 14 Bortezomib (Velcade®) : 1,3 mg/m2/d, days 1, 4, 8, et 11 Lenalidomide (Revlimid®) :25 mg/d, days 1 to 14
  Consolidation (2 months After ASCT):
  2 cycles of 21 days of Lenalidomide (Revlimid®) 25 mg/j, days 1 à 14 Bortezomib (Velcade®) 1,3 mg/m2/d, days 1, 4, 8, et 11 Dexamethasone 40 mg/j, days 1, 8 et 14
  Maintenance Phase:
  3 to 8 weeks after consolidation. Cycle length: 28 days Lenalidomide (Revlimid®) 10 mg/d until 12 months
  Other Names: Lenalidomide (REVLIMID®); Bortezomib (VELCADE®)

SUMMARY:
The purpose of this Phase 2 study is to evaluate the efficacy and safety of treatment with bortezomib, lenalidomide and dexamethasone in patients with untreated multiple myeloma. This study will evaluate whether the addition of lenalidomide to bortezomib and dexamethasone will increase the Complete Response (CR)/ very good partial response (VGPR) rate before and after High Dose Therapy (HDT) with ASCT.

DETAILED DESCRIPTION:
Patients will receive 3 induction cycles of bortezomib, lenalidomide and dexamethasone (VRD) followed by high dose melphalan and autologous stem cell transplantation. Two months after haematological recovery, patients will receive 2 consolidation cycles of VRD and maintenance therapy for 1 year with lenalidomide

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with multiple myeloma based on standard diagnostic criteria or by the new International Myeloma Foundation 2003 Diagnostic Criteria
* Subjects must have symptomatic myeloma or asymptomatic myeloma with myeloma-related organ damage
* Subjects must have measurable disease requiring systemic therapy.
* Male or female subject 18 years of age or older
* Karnofsky Performance Status score of ≥50% (Eastern Cooperative Oncology Group Performance Status score ≤2)
* Voluntary written informed consent must be given before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to therapy. They must commit to continued abstinence from heterosexual intercourse or begin 2 acceptable methods of birth control (1 highly effective method and 1 additional effective method) used at the same time, beginning at least 4 weeks before initiation of Revlimid treatment. Women must also agree to ongoing pregnancy testing
* Men must agree to not father a child and agree to use a latex condom during therapy and for 4 weeks after the last dose of study drug, even if they have had a successful vasectomy, if their partner is of childbearing potential.

Exclusion Criteria:

* Subjects must not have been treated previously with any systemic therapy for multiple myeloma. Prior treatment with corticosteroids or radiation therapy does not disqualify the subject (the maximum dose of corticosteroids should not exceed the equivalent of 160 mg of dexamethasone in a 2-week period). Two weeks must have elapsed since the date of the last radiotherapy treatment. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 2 weeks have elapsed since the last date of therapy.
* AL amylo
* ≥Grade 2 peripheral neuropathy on clinical examination within 14 days before enrollment
* Renal insufficiency (serum creatinine >2.5 mg/dL)
* Evidence of mucosal or internal bleeding and/or platelet refractory
* Platelet count <70,000 per µL
* ANC < 1000 cells/mm3
* AST or ALT greater than or equal to 2 x ULN
* Total bilirubin >3 × ULN
* Myocardial infarction within 6 months prior to enrollment according to NYHY Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Clinically relevant active infection or serious co-morbid medical conditions
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical, breast or prostate cancer
* Female subject who is pregnant or breast-feeding
* Serious medical or psychiatric illness likely to interfere with participation in study
* Uncontrolled diabetes mellitus
* Known HIV infection
* Known active hepatitis B or C viral infection
* Known intolerance to steroid therapy
* History of allergy to any of the study medications, their analogues, or excipients in the various formulations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of the best response after consolidation | 6 to 8 months after start of induction for each patient = after consolidation therapy for all patients
  Evaluate the best response achieved , according to the IMWG uniform criteria, after consolidation treatment.

SECONDARY OUTCOMES:
Response Evaluation after 3 cycles | 6 to 8 months after start of induction for each patient = after consolidation therapy for all patients
  Evaluate the complete and very good partial response rates of the combination of bortezomib, lenalidomide and dexamethasone in newly diagnosed multiple myeloma patients after 3 cycles.
Safety and tolerability : number and nature of Adverse Events | 6 to 8 months after start of induction for each patient = after consolidation therapy for all patients
  Determine the safety and tolerability of the drug combination in this patient populations.
Stem Cells Collection | 6 to 8 months after start of induction for each patient = after consolidation therapy for all patients
  Evaluate the faisability and quality of the peripheral stem cells collection.
Response After HDT-ASCT and 2 cycles | 6 to 8 months after start of induction for each patient = after consolidation therapy for all patients
  Evaluate the complete and very good partial response rates 2 months after HDT with ASCT and after 2 cycles of consolidation treatment.
Progression Free Survival | 6 to 8 months after start of induction for each patient = after consolidation therapy for all patients
  Evaluate the progression free survival, the overall survival, time to progression and duration of response.

CONTACTS AND LOCATIONS:
Overall Officials: Michel ATTAL, MD, Principal Investigator — University Hospital of Toulouse
Locations (9):
- France (9):
  - Centre François Baclesse, Caen
  - University Hospital of Dijon, Hôpital des Enfants, Dijon
  - University Hospital of Grenoble, Hôpital A.Michallon, BP 217 X, Grenoble
  - University Hospital Of Lille, Hôpital Claude Huriez, Lille
  - Institut Paoli Calmette, Marseille
  - University Hospital of Bordeaux, "Hôpital du Haut Lévêque ", Pessac
  - University Hospital of Toulouse, Purpan, Toulouse
  - Hôpital Bretonneau, Tours, Tours
  - Hôpitaux de Brabois Nancy, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Roussel M, Lauwers-Cances V, Robillard N, Hulin C, Leleu X, Benboubker L, Marit G, Moreau P, Pegourie B, Caillot D, Fruchart C, Stoppa AM, Gentil C, Wuilleme S, Huynh A, Hebraud B, Corre J, Chretien ML, Facon T, Avet-Loiseau H, Attal M. Front-line transplantation program with lenalidomide, bortezomib, and dexamethasone combination as induction and consolidation followed by lenalidomide maintenance in patients with multiple myeloma: a phase II study by the Intergroupe Francophone du Myelome. J Clin Oncol. 2014 Sep 1;32(25):2712-7. doi: 10.1200/JCO.2013.54.8164. Epub 2014 Jul 14. PMID 25024076